CLINICAL TRIAL: NCT04991493
Title: Effect of Tramadol on Postoperative Sore Throat in Thyroid Surgery Under General Anesthesia With Endotracheal Intubation: A Randomized Controlled Trial
Brief Title: Effect of Tramadol on Postoperative Sore Throat After General Anesthesia
Status: Recruiting | Phase: Phase 4 | Type: Interventional
Sponsor: Affiliated Cancer Hospital of Shantou University Medical College (Other)
Responsible Party: Principal Investigator, zegeng su, Attending doctor/ Master of medicine, Affiliated Cancer Hospital of Shantou University Medical College
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Prevention
Other Study IDs: QPOST
Record Dates: First submitted 2021-07-27; First posted 2021-08-05 (Actual); Last update posted 2024-05-13 (Actual); Status verified 2024-05

CONDITIONS: Post-operative Sore Throat; Intubation Intratracheal; Thyroid Surgery
Keywords: Tramadol; Post-operative Sore Throat; Intubation, Intratracheal; thyroid surgery
MeSH Terms: interventions — Tramadol; Saline Solution

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Masking Description: The anesthesia provider will be blinded to the intervention group allocation. All patients will be blinded. The primary investigator will be blinded. The resident researcher who will be the outcome assessor will also be blinded. The care provider will be blinded.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: Yes

ARMS (3):
- Placebo group (Placebo Comparator): 5ml normal saline was injected intravenously 15 minutes before anesthesia and 5ml normal saline was injected intravenously when the incision was washed and sutured.
  Interventions: Other: Normal Saline
- pre-tramadol group (Experimental): 5ml of tramadol containing 1mg / kg was injected intravenously 15 minutes before anesthesia and 5ml of normal saline was injected intravenously when the incision was washed and sutured.
  Interventions: Drug: Tramadol hydrochloride
- post-tramadol group (Active Comparator): 5ml of normal saline was injected intravenously 15 minutes before anesthesia and 5ml of tramadol containing 1mg / kg was injected intravenously when the incision was washed and sutured.
  Interventions: Drug: Tramadol hydrochloride

INTERVENTIONS:
Drug: Tramadol hydrochloride — pre-tramadol group: 1mg/kg of tramadol will be intravenously injected 15 minutes before anesthesia.
  post-tramadol group: 1mg/kg of tramadol will be intravenously injected when the incision was washed and sutured.
  Other Names: Tramadol
  Arms: post-tramadol group; pre-tramadol group
Other: Normal Saline — pre-tramadol group: Normal Saline will be injected intravenously when the incision was washed and sutured.
  post-tramadol group: Normal Saline will be injected intravenously 15 minutes before anesthesia.
  Arms: Placebo group

SUMMARY:
Post operative sore throat after general anesthesia with endotracheal intubation is a common problem causing dissatisfaction and discomfort to the patients. The investigators want to study the effect of tramadol on postoperative sore throat in general anesthesia with endotracheal intubation.

DETAILED DESCRIPTION:
Design: A prospective, randomized, controlled study. Setting: Single-center university hospital. Participants: The study included 168 patients undergoing thyroid surgery under general anesthesia with endotracheal intubation.

Interventions: The patients were allocated randomly into the following 3 groups: the control group: patients will be injected intravenously 5ml of normal saline 15 minutes before anesthesia and another 5ml of normal saline was injected intravenously when the incision was washed and sutured；the pre-tramadol group: patients will be injected intravenously 5ml of tramadol (1mg / kg) 15 minutes before anesthesia and 5ml of normal saline was injected intravenously when the incision was washed and sutured. the post-tramadol group: patients will be injected intravenously 5ml of normal saline 15 minutes before anesthesia and 5ml of tramadol (1mg / kg) was injected intravenously when the incision was washed and sutured. Postoperatively, all patients will receive standard treatment.

ELIGIBILITY:
Inclusion Criteria:

- Female with American Society of Anesthesiologists (ASA) physical status I-II; Elective thyroidectomy(non-endoscopic) with endotracheal intubation; The patient signed the consent form.

Exclusion Criteria:

- History of thyroid surgery A history of preoperative sore throat; Pregnancy; Retrosternal goiter; Thyroid tumor invading trachea need trachea reconstruction; Potentially difficult airway; Clinical diagnosis of chronic sore throat; Clinical diagnosis of psychosis; Tracheotomy after operation； Transfer to intensive care unit after operation； Contraindications to tramadol； Body mass index (BMI) > 30kg/m^2.

Ages: 18 Years to 65 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Gender Based: Yes — Gender is one of the independent factors affecting postoperative sore throat. To reduce the bias from gender, we only considered female patients.
Enrollment: 168 (Estimated)
Dates: Start 2021-09-10 (Actual); Primary Completion 2023-11-01 (Actual); Study Completion 2024-07 (Estimated)

PRIMARY OUTCOMES:
The Incidence of Post-operative sore throat | 24 hours following extubation of endotracheal tube
  The incidence of postoperative sore throat at 24 hours after extubation.

SECONDARY OUTCOMES:
The Incidence of Post-operative sore throat | 30 Minutes following extubation of endotracheal tube
  The incidence of postoperative sore throat at 0 hours and 4 hours after extubation.
The Incidence of Post-operative sore throat | 4 hours following extubation of endotracheal tube
  The incidence of postoperative sore throat at 0 hours and 4 hours after extubation.
The severity of Post-Operative Sore Throat | 30 Minutes ，4 hours and 24 hours following extubation of endotracheal tube
  Assessment of severity of postoperative sorethroat using scoring system, 0-No sore throat at any time since the extubation,1- Minimal sore throat,2- Moderate sore throat,3- Severe sore throat
The incidence of of postoperative hoarseness. | 30 Minutes ，4 hours and 24 hours following extubation of endotracheal tube
  The incidence of of postoperative hoarseness at 0 hours，4 hours and 24 hours after extubation.
The severity of postoperative hoarseness | 30 Minutes ，4 hours and 24 hours following extubation of endotracheal tube
  Assessment of postoperative hoarseness using scoring system,0- No evidence of hoarseness at any time since the extubation,1-No evidence of hoarseness at the time of interview,2-Hoarseness at the time of interview noted by patient only, 3- Hoarseness that is easily noted at the time of interview

CONTACTS AND LOCATIONS:
Overall Officials: zegeng su, master, Principal Investigator — Affiliated Cancer Hospital of Shantou University Medical College Medical
Locations (1):
- Affiliated Cancer Hospital of Shantou University Medical College Medical, Shantou, Guangdong, China

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Hu B, Bao R, Wang X, Liu S, Tao T, Xie Q, Yu X, Li J, Bo L, Deng X. The size of endotracheal tube and sore throat after surgery: a systematic review and meta-analysis. PLoS One. 2013 Oct 4;8(10):e74467. doi: 10.1371/journal.pone.0074467. eCollection 2013. PMID 24124452
- [Background] El-Boghdadly K, Bailey CR, Wiles MD. Postoperative sore throat: a systematic review. Anaesthesia. 2016 Jun;71(6):706-17. doi: 10.1111/anae.13438. Epub 2016 Mar 28. PMID 27158989
- [Background] Tekelioglu UY, Apuhan T, Akkaya A, Demirhan A, Yildiz I, Simsek T, Gok U, Kocoglu H. Comparison of topical tramadol and ketamine in pain treatment after tonsillectomy. Paediatr Anaesth. 2013 Jun;23(6):496-501. doi: 10.1111/pan.12148. Epub 2013 Mar 23. PMID 23521170
- [Background] Lin BF, Ju DT, Cherng CH, Hung NK, Yeh CC, Chan SM, Wu CT. Comparison between intraoperative fentanyl and tramadol to improve quality of emergence. J Neurosurg Anesthesiol. 2012 Apr;24(2):127-32. doi: 10.1097/ANA.0b013e31823c4a24. PMID 22089326